CLINICAL TRIAL: NCT04483479
Title: A Multicenter, Non-Randomized, Open-Label Study to Evaluate the Safety and Efficacy of Orally Administered ENT-01 in Improving Constipation and Neurologic Symptoms in Patients With Parkinson's Disease and Constipation Over a 14-week Period
Brief Title: Orally Administered ENT-01 for Parkinson's Disease-Related Constipation Follow-on Safety "Roll-over" Study (Rollover)
Acronym: Rollover
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment/retention due to the pandemic. Data was not analyzed due to early termination.
Sponsor: Enterin Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENT-01-2b-20-02
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Constipation
MeSH Terms: conditions — Parkinson Disease; Constipation

STUDY DESIGN:
Intervention Model Description: This is a Phase 2b, non-randomized, open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Treatment (Experimental): Orally Administered ENT-01 25mg Tablet Once Daily (Dose dependent on ENT-01-030 dose level stratification)
  Interventions: Drug: Active Investigational Treatment ENT-01

INTERVENTIONS:
Drug: Active Investigational Treatment ENT-01 — ENT-01 will be administered in tablet form, once daily in escalating doses followed by a fixed-dose for 12 weeks.
  Other Names: ENT-01

SUMMARY:
This study will be conducted as an open-label safety follow-on to a multi-center, double-blind, randomized study. All subjects who participated in the randomized study will be offered participation in this unblinded, single-arm, safety study. Approximately 50 subjects will be entered into the study and ENT-01 will be administered daily in escalating doses followed by a fixed dose for 12 weeks. Each subject will participate for approximately 20 weeks; dosing duration will be approximately 14 weeks.

DETAILED DESCRIPTION:
The study will be conducted on an out-patient or in-patient basis with visits performed at the screening visit, at 6 and 12 weeks, and at the end of the 6th week of the wash-out period (end of study).

The dose escalation period will last up to 20 days, the fixed dose period will last 12 weeks, and the wash-out period will last 6 weeks.

Subjects will begin dosing at the same dose level they were stratified to in the ENT-01-030 randomized study (i.e., starting at either 3 tablets or 6 tablets,) and escalate up to a pro-kinetic dose or a maximum dose of 250mg.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects who participated in the randomized study ENT-01-030 (KARMET Stage 2 Extension subjects) and who completed the dosing period.
2. Subjects aged 30-90 years at the time of screening for the ENT-01-030 study, both genders
3. Subjects must provide informed consent and be willing and able to comply with study procedures.
4. Subjects must be able to read, understand, and accurately record data into the diary to guarantee full participation in the study.
5. Female subjects must have negative serum or urine pregnancy tests and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. A vasectomized partner will be allowed as one in conjunction with another single-barrier method.
6. Female subjects unable to bear children must have this documented in the CRF (i.e., tubal ligation, hysterectomy, or postmenopausal [defined as a minimum of one year since the last menstrual period]). Post-menopausal status will be confirmed by follicle stimulating hormone (FSH) in women less than 60 years of age.

Exclusion Criteria:

1. Unable or unwilling to provide informed consent or to comply with study procedures.
2. Unable to withdraw proton pump inhibitors.
3. Unable or unwilling to withdraw from laxatives, opiates, clonazepam, or any medications which may cause constipation 2 weeks prior to the dose adjustment period and throughout the rest of the study.
4. Diagnosis of secondary constipation beyond that of Parkinson's disease.
5. A compromised gastrointestinal system which includes:

   * Structural, metabolic, or functional GI diseases or disorders.
   * Acute GI illness within 2 weeks of the screening visit.
   * History of major GI surgery within 30 days of the screening visit (a history of cholecystectomy, polypectomy, hernia repair or appendicectomy are not exclusionary as long as they were performed more than 30 days before the screening visit).
6. Neurological disorder other than Parkinson's disease that in the opinion of the investigator might interfere with the conduct of the study.
7. On treatment with intra-jejunal dopamine or carbidopa/levodopa (i.e. Duopa).
8. Subjects starting a new Parkinson's disease medication or modifying an existing medication within 2 weeks prior to enrollment.
9. Unable to maintain a stable diet regimen.
10. Subjects with a cognitive impairment that preclude them from understanding the informed consent.
11. Subjects placed under legal guardianship.
12. History of excessive alcohol use or substance abuse.
13. Any clinically significant abnormalities on screening laboratories or physical examination requiring further evaluation or treatment.
14. Females who are pregnant or breastfeeding.
15. Subject or caregiver unable to administer daily oral dosing of study drug.
16. Participation in a non-Enterin investigational drug trial within the month prior to dosing in the present study.
17. Any other reason, which in the opinion of the investigator would confound proper interpretation of the study.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zasloff, MD, PhD, Study Chair — Enterin Inc.; Denise Barbut, MD, FRCP, Study Director — Enterin Inc.
Locations (18):
- United States (18):
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - SC3 Research - Pasadena, Pasadena, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Georgetown Universtiy, Department of Neurology, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Parkinson's Disease Treatment Center of SWFL, Port Charlotte, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - USF Health Byrd Parkinson's Disease Movement Disorders Center of Excellence, Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Penn State University, Hershey, Pennsylvania
  - Evergreen Health - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - University Physicians & Surgeons, Inc. dba Marshall Health, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment
Started | 27
Completed | 12
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Active Treatment
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27
BMI [Mean (Standard Deviation); unit: KG/m^2] | 26.7 (4.63)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Description: Number of participants with Treatment Related Adverse Events
Time Frame: Through study treatment and completion up to 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment
Number analyzed (Participants) | 27
Participants | 23

2. Primary Outcome: Number of Participants With Treatment Related Recurrent Vomiting
Description: The number of participants with treatment related episodes of recurrent vomiting defined as 3-5 episodes of vomiting within 24 hours
Time Frame: Through study treatment and completion up to 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment
Number analyzed (Participants) | 27
Participants | 5

3. Primary Outcome: Number of Participants With Treatment Related Recurrent Diarrhea
Description: The number of participants with treatment related episodes of recurrent diarrhea defined as 7 episodes of diarrhea within 24 hours for 2 consecutive days
Time Frame: Through study treatment and completion up to 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment
Number analyzed (Participants) | 27
Participants | 8

4. Primary Outcome: Number of Participants With Treatment Related Dizziness
Description: The number of participants with treatment related episodes of dizziness defined as lightheadedness or fainting on rising from lying to sitting or standing and severe enough to require non-urgent medical intervention within 24 hours
Time Frame: Through study treatment and completion up to 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment
Number analyzed (Participants) | 27
Participants | 8

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 24/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment (N=27)
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 8
Tremors (Nervous system disorders) | 2
Weight Decreased (Investigations) | 2
Dizziness (Vascular disorders) | 8

LIMITATIONS AND CAVEATS:
Study was terminated early due to poor recruitment/retention due to the pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT04483479/Prot_SAP_001.pdf